CLINICAL TRIAL: NCT07001397
Title: Study on the Short-term Efficacy and Safety of Recombinant Human Thrombopoietin Combined With Immunosuppressant Sequential Eltrombopag Ethanolamine Dry Suspension in the Treatment of SAA/TD-NSAA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPO-2024-016
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Aplastic Anemias
Keywords: Aplastic anemia; rhTPO; EPAG-pfos
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rhTPO+IST+EPAG-pfos (Active Comparator)
  Interventions: Drug: EPAG-pfos

INTERVENTIONS:
Drug: EPAG-pfos — The initial dose of EPAG-pfos is 150mg/d orally. The dose is adjusted according to hematological indicators, with a maximum dose of 150mg/d until hematological remission is achieved

SUMMARY:
The study included adult patients ≥18 years old with SAA and TD-NSAA who had no HLA-matched sibling donors or were not suitable for first-line allogeneic hematopoietic stem cell transplantation due to age, complications, patient wishes, etc. After admission, they were treated with standard IST combined with rhTPO for at least 28 days. After discharge, the sequential treatment of EPAG-PFOS (with an initial dose of 150mg/d) was continued for 2 months (8 weeks), and the follow-up was conducted until the 6th month (24 weeks). It was compared with the historical cohort previously treated with IST combined with EPAG to explore the short-term efficacy and safety of this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender not limited;
2. Patients diagnosed with aplastic anemia (AA) through blood routine, bone marrow puncture, bone marrow biopsy and excluded examinations, and determined as SAA or TD-NSAA according to the Camitta criteria;
3. Those who have not received treatment with immunosuppressants (such as cyclosporine, tacrolimus, ATG, etc.);
4. The patient has no HLA-matched sibling donor or is not suitable for first-line allogeneic hematopoietic stem cell transplantation due to reasons such as age, complications, or the patient's wishes.
5. Before treatment, the total bilirubin (TBIL) of the patient was less than 1.5 times the upper limit of normal value (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were less than 3 times the ULN, and serum creatinine was less than 1.5 times the ULN.
6. ECOG score ≤2 points;
7. Voluntarily join this study, sign the informed consent form, have good compliance and be willing to cooperate with regular follow-up for therapeutic effect evaluation and side effect monitoring;

Exclusion Criteria:

1. Pregnant or lactating patients;
2. Have a history of any arterial or venous thrombosis (including stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism) within half a year before enrollment and have at least two of the following risk factors: Hormone replacement therapy, oral contraceptives (including estrogen), smoking, diabetes, hypercholesterolemia, drug-controlled hypertension, hereditary coagulation disorders;
3. Patients with severe cardiovascular diseases (such as NYHA Cardiac Function Score grade III-IV) within half a year before enrollment, known arrhythmias that increase the risk of thromboembolism such as atrial fibrillation, after coronary stent implantation, angioplasty, and after coronary artery bypass grafting;
4. Combined with malignant tumors that seriously affect survival;
5. Within 2 weeks after the start of the study until the end of the study, continuous drug treatment (including but not limited to aspirin, clopidogrel and/or non-steroidal anti-inflammatory drugs NSAIDs) or anticoagulant treatment that affects platelet function for more than 3 days;
6. Currently, there is a severe or difficult-to-control infection (CTC AE level 2 infection);
7. Bone marrow biopsy within 4 weeks before the administration of the first dose of the study indicates the presence of primary diseases other than SAA that can cause thrombocytopenia (such as primary myelodysplastic syndrome (MDS), congenital bone marrow failure diseases (such as Fanconi anemia, congenital keratosis, etc.) Or accompanied by obvious paroxysmal nocturnal hemoglobinuria (PNH) clones (> 50%) and AA with clinical and biochemical indicators of hemolysis; And the researcher judged that the subject was not suitable to participate in this study.
8. All laboratory or clinical evidence of HIV infection, previous clinical history of hepatitis C, previous hepatitis B infection, or active hepatitis at the time of screening. Laboratory tests during the screening period indicated hepatitis C infection or hepatitis B infection. (Defined as a positive HBsAg test. Additionally, if the HBsAg test is negative but HBcAb is positive, regardless of the status of HBsAb, HBV DNA testing is required. If it is positive, the subject should be excluded.)
9. Chronic liver disease-related AA (hepatitis disease-related AA, liver cirrhosis, etc.);
10. Had received treatment with TPO or TPO receptor agonists (TPO-RAS, including but not limited to eltrombopag, romisetine, avatrombopag, heltrombopag, rutrombopag, etc.) before screening;
11. Suffer from severe autoimmune diseases or immunodeficiency diseases;
12. Suffer from serious mental disorders;
13. Patients who the researchers consider unsuitable to participate in this trial, such as those with any other medical, social or psychological factors that may affect safety or compliance with the research procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2026-03-23 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 1 month, 3 month

IPD SHARING:
Plan to Share IPD: No